CLINICAL TRIAL: NCT05645627
Title: A Phase Ⅲ, Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of IBI112 in Different Dose Regimens for the Treatment of Subjects With Moderate-to-severe Plaque Psoriasis
Brief Title: A Study to Evaluate IBI112 in the Treatment of Psoriasis With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI112A301
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Placebo Comparator): Participants receive placebo through week 16,placebo participants will cross over to receive IBI112 through week 48
  Interventions: Drug: placebo /IBI112
- Group 2 (Experimental): Participants receive Dose 1 IBI112 through week 16 ,and then will receive Dose 2 IBI112 through week 48
  Interventions: Drug: IBI112
- Group 3 (Experimental): Participants receive Dose 1 IBI112 through week 16 ,and then will receive Dose 3 IBI112 through week 48
  Interventions: Drug: IBI112

INTERVENTIONS:
Drug: IBI112 — IBI112 by subcutaneous injection through week 16 ,and then will receive Dose 3 IBI112 by subcutaneous injection through week 48
  Arms: Group 2
Drug: placebo /IBI112 — placebo by subcutaneous injection cross over IBI112 by subcutaneous injection at week 16 through week 48
  Arms: Group 1
Drug: IBI112 — IBI112 by subcutaneous injection through week 16 ,and then will receive Dose 3 IBI112 by subcutaneous injection through week 48
  Arms: Group 3

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of IBI112 in the treatment of participants with moderate to severe plaque-type psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of plaque-type psoriasis with or without psoriatic arthritis for at least 6 months prior to first administration of any study agent
2. Must be a candidate for phototherapy or systemic treatment for psoriasis (either new to treatment or having had previous treatment)

Exclusion Criteria:

1. History of or current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease
2. Participant has history of erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new onset guttate psoriasis
3. Has received any therapeutic agent directly targeted to IL-17within 6 months of the first administration of study agent
4. Has received any therapeutic agent directly targeted toTNF-a within 3 months of the first administration of study agent
5. Has received any conventional therapeutic agent within 1 months of the first administration of study agent
6. Has received any topic therapeutic agent within 2 weeks of the first administration of study agent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving Psoriasis Area and severity index(PASI) 90 at week 16 | Week 16
  PASI 90 is defined as at least a 90% reduction in PASI relative to baseline
Percentage of patients achieving an static Physician's Global Assessment (sPGA) Score of Cleared (0) or Minimal (1) at Week 16 | Week 16
  sPGA of psoriasis is used to determine the participant's psoriasis lesions overall at a given time point. sPGA score ranges from 0-4,0=cleared, 1= minimal ,2=mild, 3= moderate, 4= marked, 5= severe

SECONDARY OUTCOMES:
Percentage of patients achieving Psoriasis Area and severity index(PASI) 75 at week 16 | Week 16
  PASI 75 is defined as at least a 75% reduction in PASI relative to baseline
Percentage of patients achieving Psoriasis Area and severity index(PASI) 100 at week 16 | Week 16
  PASI 100 is defined as at least a 100% reduction in PASI relative to baseline
Percentage of patients achieving an static Physician's Global Assessment (sPGA) Score of Cleared (0) at Week 16 | Week 16
  sPGA of psoriasis is used to determine the participant's psoriasis lesions overall at a given time point. sPGA score ranges from 0-4,0=cleared, 1= minimal ,2=mild, 3= moderate, 4= marked, 5= severe
Change from Baseline in Dermatology life quality index(DLQI) at week 16 | Week 16
  The DLQI is a 10-item questionnaire that measures the impact of skin disease on participant's quality of life
Percentage of patients achieving Psoriasis Area and severity index(PASI) 90 at week 52 | Week 52
  PASI 90 is defined as at least a 90% reduction in PASI relative to baseline
Percentage of patients achieving an static Physician's Global Assessment (sPGA) Score of Cleared (0) or Minimal (1) at Week 52 | Week 52
  sPGA of psoriasis is used to determine the participant's psoriasis lesions overall at a given time point. sPGA score ranges from 0-4,0=cleared, 1= minimal ,2=mild, 3= moderate, 4= marked, 5= severe
Percentage of patients achieving Psoriasis Area and severity index(PASI) 75 at week 52 | Week 52
  PASI 75 is defined as at least a 75% reduction in PASI relative to baseline
Percentage of patients achieving Psoriasis Area and severity index(PASI) 100 at week 52 | Week 52
  PASI 100 is defined as at least a 100% reduction in PASI relative to baseline
Percentage of patients achieving an static Physician's Global Assessment (sPGA) Score of Cleared (0) at Week 52 | Week 52
  sPGA of psoriasis is used to determine the participant's psoriasis lesions overall at a given time point. sPGA score ranges from 0-4,0=cleared, 1= minimal ,2=mild, 3= moderate, 4= marked, 5= severe
Change from Baseline in Dermatology life quality index(DLQI) at week 52 | Week 52
  The DLQI is a 10-item questionnaire that measures the impact of skin disease on participant's quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality, China